CLINICAL TRIAL: NCT03904017
Title: The Role of Hyperoxia in the Emergency Department Treatment of Acute Ischemic Stroke
Brief Title: The Role of Hyperoxia in Acute Ischemic Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to enroll
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-0486
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperoxia (Experimental): Will receive 15liters per minute supplemental oxygen via a partial non-rebreather facemask.
  Interventions: Other: Oxygen
- Placebo (Placebo Comparator): will receive 15liters per minute medical air via a partial non-rebreather facemask.
  Interventions: Other: placebo

INTERVENTIONS:
Other: Oxygen — 100% Oxygen air
  Arms: Hyperoxia
Other: placebo — medical air
  Arms: Placebo

SUMMARY:
This study is being conducted to evaluate the potential therapeutic role of hyperoxia when applied in the immediate ischemic period following a stroke in the controlled Emergency Department setting. The study will evaluate the effects of hyperoxia in stroke patients on the production of markers of free radical damage and inflammatory markers associated with hyperoxic lung injury.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form from patient or legal authorized representative (LAR)
2. Subject or LAR stated willingness to comply with all study procedures and availability for the duration of the study
3. Males and females (of unlikely childbearing capacity) aged over 18 years.
4. Exhibiting signs and physical examination findings suggestive of an acute ischemic infarction (either a or b)

   1. A target mismatch profile of CT-perfusion or MRI determined by RAPID automated software to have a ratio of PWITmax>6 lesion volume/DWI lesion volume >1.2 and an NIHSS >/=1
   2. A RAPID automated software calculated non-contrast CT-head ASPECT score of 10 and LKW ≤12 hours (in patients with symptoms discovered upon waking, the LKW is defined at the midpoint between going to sleep and awakening based on previous studies that suggest most strokes during sleep occur close to awakening)
5. Normoxic; a pulse oximetry of 94% or greater at time of screening without the use of supplemental oxygen

Exclusion Criteria:

1. Current use of supplemental oxygen
2. Prisoner
3. Documented blood glucose <70mg/dL
4. Concurrent treatment with another investigational drug or other intervention
5. Documented history of any of the following chronic respiratory illness that require pulmonary vasodilators or supplemental oxygen at baseline: Chronic Obstructive Pulmonary Disorder (COPD), Emphysema, Interstitial Lung Disease, Restrictive Lung Disease, Pulmonary Hypertension
6. Documented history of any of the following autoimmune diseases: systemic lupus erythematosus, rheumatoid arthritis, scleroderma, primary biliary cholangitis, multiple sclerosis, inflammatory bowel disease
7. Currently being treated for an acute myocardial infarction and/or decompensated heart failure at the onset of initial ED presentation as reported by the ED provider
8. Plans for treatment with either IV tPA (alteplase) or endovascular therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Colorado, Aurora, Colorado
  - University of Colorado Hospital - Memorial Central, Colorado Springs, Colorado

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hyperoxia | Placebo
Started | 3 | 10
Completed | 3 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hyperoxia | Placebo | Total
Number analyzed (Participants) | 3 | 10 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 2 | 7 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (17.4) | 71.6 (14.3) | 68.9 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 6 | 6
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 10 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 2 | 9 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 10 | 13

OUTCOME MEASURES:

1. Primary Outcome: Mean Time to Randomization and Initiation of Intervention
Description: Patient arrival to the emergency department will be documented and recorded. They will be screened for participation by study personnel. Once consented and randomized, the time of initiation of intervention will be recorded. The mean time from emergency department presentation to initiation of therapy will be determined.
Time Frame: baseline
Population: The time from ED arrival to initiation of treatment arm was measured in minutes for 3 patients receiving hyperoxia and 10 patients receiving placebo
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Hyperoxia | Placebo
Number analyzed (Participants) | 3 | 10
minutes | 96.7 (27.3) | 75.1 (14.8)

2. Secondary Outcome: Mean Ratio of the Volume of Initial Hypoperfused Tissue to Final Infarct Volume
Description: The total area of hypoperfused brain tissue on initial imaging will be compared to the final infarct volume. This ratio of hypoperfused to final infarct volume will be compared between treatment groups.
Time Frame: one week
Population: Subjects (3 hyperoxia and 6 placebo) who were able to complete the MRI within one week had the volume of the total hypoperfused brain tissue and the final infarct volume measured using RAPID automated software.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Hyperoxia | Placebo
Number analyzed (Participants) | 3 | 6
ratio | 2.17 (0.69) | 7.76 (10.7)

3. Secondary Outcome: Change in Mean NIHSS
Description: National Institute of Health Stroke Scale (NIHSS) score will be measured at presentation and 24-hours after intervention. The change in NIHSS from presentation to 24-hours will be compared between groups. The NIHSS score is a range of scores from 0-42 with higher scores indicating a more severe stroke and disability.
Time Frame: baseline to 24-hours
Population: The change in NIHSS from baseline to 24 hours was calculated for 3 hyperoxia and 10 placebo subjects. The mean and standard deviation for both groups was calculated
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hyperoxia | Placebo
Number analyzed (Participants) | 3 | 10
score on a scale | 2 (0) | 1.2 (3.1)

ADVERSE EVENTS:
Time Frame: Subjects were monitored for adverse events during the 24hours that they were under study observation. A 90-day modified Rankin was collected and any deaths at this time were noted.
Arm/Group | Hyperoxia | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/10
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/10
Other Adverse Events (participants affected / at risk) | 0/3 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT03904017/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT03904017/ICF_001.pdf